CLINICAL TRIAL: NCT02190422
Title: Effect of Assisted Reproductive Technology on Cardiac Development in Childhood Assessed by Echocardiography
Acronym: Heart and ART
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, Principal Investigator, Nanjing Medical University
Other Study IDs: 2012CB944902
Record Dates: First submitted 2014-07-10; First posted 2014-07-15 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Assisted Reproductive Technology
Keywords: reproductive technologies, assisted; echocardiography; cardiology; pediatrics
MeSH Terms: conditions — Helping Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Assisted reproductive technology (ART) has extensively allowed pregnancy for infertile couples. However, the long-term effect of ART exposure on cardiovascular development and potential association with ART procedure and parental factors is confused. The aim is to shed more light on the pattern and extent of cardiovascular developmental alteration among ART children and its association with potential confounders.

DETAILED DESCRIPTION:
A historic cohort study was designed with prospective follow-up of ART children conceived in the Clinical Centre of Reproductive Medicine (CCRM) and born in Maternal-Fetal Medicine Unit (MFMU) of First Affiliated Hospital of Nanjing Medical University (FAHNMU) from 1 January 2002 to 31 December 2012.

The present design is a prospective single-center study in FAHNMU. ART group will be recruited by a non-random, consecutive sample on the basis of the unique personal identification number assigned to ART children conceived in CCRM and born in MFMU.

The controls will be recruited by a non-random, consecutive sample on the basis of the spontaneous conception population attending the MFMU of FAHNMU during the same period as ART group for prenatal screening and subsequent delivery considering their age.

ELIGIBILITY:
Inclusion Criteria:

* the capability of complete examination of transthoracic echocardiography
* the absence of complex cardiac malformations and systematic diseases.

Exclusion Criteria:

* the presence of a history of systemic diseases, frequent arrhythmias, and critical acquired heart diseases,
* the presence of the background of familiar cardiomyopathy in their family,
* limited acquisitions of echocardiographic imaging
* poor image quality for assessment.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: ART group will be ART children conceived in Clinical Centre of Reproductive Medicine and born in Maternal-Fetal Medicine Unit (MFMU). The controls will be the spontaneous conception children born in the MFMU during the same period as ART group for prenatal screening and subsequent delivery.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
cardiovascular geometric morphology between controls and ART children | participants will be followed for the duration of hospital stay, an expected average of 3 weeks
  Left ventricular end-diastolic diameters (LVDD) and end-systolic diameters (LVSD) will be measured by M-mode echocardiography at the para-sternal long-axis views. LV end-diastolic volume (LVEDV) and end-systolic volume(LVESV) will be calculated by 2D echocardiography from the apical four-chamber view using the modiﬁed Simpson's rule. Aorta diameters (AOD) and left atrial diameters (LAD) will be measured by 2D echocardiography at the para-sternal long-axis views. Left and right coronary artery will be measured by 2D echocardiography at the short-axis views. The interventricular septum thickness (IVST) and the left ventricular posterior wall thickness (LVPWT) will be measured by M mode from a para-sternal long-axis view. Left ventricular relative wall thickness (LVRWT) will be calculated the following equation: (IVST+PWT)/ LVDD.

SECONDARY OUTCOMES:
cardiac function between controls and ART children | participants will be followed for the duration of hospital stay, an expected average of 3 weeks
  LV shortening fraction will be calculated from internal ventricular diameters obtained from a para-sternal long-axis view by M mode using the following equation: (end-diastolic diameter-end-systolic diameter)/end-diastolic diameter. LV stroke volumes will be calculated as follows: π/4×(aortic valve diameter)2×(aortic artery systolic flow velocity-time integral). Left ejection fraction will be calculated as follows: (end-diastolic volume-end-systolic volume)/end-diastolic volume. Left cardiac outputs will be calculated as stroke volume times heart rate. Left cardiac index will be normalized as cardiac outputs/ BSA.

CONTACTS AND LOCATIONS:
Locations (1):
- Philips Ultrasound, Nanjing, Jiangsu, China

REFERENCES:
- [Result] Liu H, Zhang Y, Gu HT, Feng QL, Liu JY, Zhou J, Yan F. Association between assisted reproductive technology and cardiac alteration at age 5 years. JAMA Pediatr. 2015 Jun;169(6):603-5. doi: 10.1001/jamapediatrics.2015.0214. No abstract available. PMID 25915111
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Association+between+assisted+reproductive+technology+and+cardiac+alteration+at+age+5+years.